CLINICAL TRIAL: NCT00395889
Title: Effects of a 6-month Outpatient Rehabilitation Program Including Structured Exercise Training on Participation in Physical Activities in Daily Life in Lung Transplant Recipients
Brief Title: Physical Activities in Daily Life After Lung Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other); International Society for Heart and Lung Transplantation (Other)
Responsible Party: Daniel Langer, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ML3782
Record Dates: First submitted 2006-11-03; First posted 2006-11-06 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: Lung Transplantation
Keywords: Lung Transplantation; Physical Activities in Daily Life; Pulmonary Rehabilitation; Functional Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rehabilitation + Lifestyle Counseling (Experimental): Multicomponent Pulmonary Rehabilitation Program including structured exercise training
  Interventions: Procedure: Rehabilitation including structured exercise training
- Lifestyle Counseling (Active Comparator)
  Interventions: Procedure: Physical Activity Counseling

INTERVENTIONS:
Procedure: Rehabilitation including structured exercise training — Rehabilitation of at least 8 weeks, for at least twice/week. This group will also receive the exercise counseling as a part of the rehabilitation program.
  Other Names: Physical Activity Counseling; Pulmonary Rehabilitation
  Arms: Rehabilitation + Lifestyle Counseling
Procedure: Physical Activity Counseling — Six exercise counseling sessions will be carried out during a 6-month period. This group will only receive the counseling and no formal structured exercise training sessions.
  Arms: Lifestyle Counseling

SUMMARY:
The purpose of this study is to compare participation in physical activities in daily life and functional outcomes of lung transplant recipients attending a six-month multicomponent rehabilitation program including exercise training against others receiving only instructions on how to increase their participation in physical activities in daily life.

DETAILED DESCRIPTION:
At present it is not clear whether it is necessary for lung transplant recipients to participate in a rehabilitation program including structured exercise training. Observations from available studies suggest that exercise capacity and health status improve following transplantation but remain impaired when compared with values of age-matched reference groups. No differences were found between participants of rehabilitation programs and patients engaging in usual daily activities. One should be cautious however to draw definite conclusions from these findings since they rest solely on results of cross-sectional investigations or single group studies. No information on functional outcomes such as participation in physical activities in daily life is currently available in lung transplant recipients. In order to answer the question if it is necessary for lung transplant recipients to participate in an outpatient rehabilitation program including structured exercise training it is our purpose to conduct a randomized clinical trial to investigate the effects of pulmonary rehabilitation after transplantation.

* Interventions: Both groups will receive counseling to engage in regular physical activity. Patients in the intervention group will additionally follow a standardized outpatient pulmonary rehabilitation program for 6 months starting immediately after discharge from hospital.
* Hypothesis: Our alternative hypothesis is that intensive post transplant rehabilitation does enhance improvements in functional status and participation in physical activities in daily life after transplantation.
* Outcomes: Participation in physical activities in daily life will be the primary outcome. Physical component summary scale of the SF-36, exercise capacity and peripheral muscle function will be secondary outcomes. Outcomes will be assessed on discharge from the hospital and again three, six and twelve months after discharge.
* Treatment failure: Patients in the control group receiving only counseling will be allowed to discontinue the assigned treatment and will receive respiratory rehabilitation including exercise training if functional outcomes do not improve or participation in physical activities in daily life does not increase within the first three months of the intervention period. The treatment groups will be compared both as randomized (according to intention to treat) and with crossover cases excluded.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of single or double lung transplants

Exclusion Criteria:

* Recipients of multiple organ transplants
* Patients scheduled for retransplantation
* Patients not leaving hospital within 6 weeks after surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Participation in Physical Activities in Daily Life | One year

SECONDARY OUTCOMES:
Health Status (SF-36) | One year
Exercise Capacity | One year
Peripheral Muscle Function | One year
Psychological Functioning | One year

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Langer, MSc, Principal Investigator — KU-Leuven, Faculty of Movement and Rehabilitation Sciences; Rik Gosselink, PhD, Study Chair — KU-Leuven, Faculty of Movement and Rehabilitation Sciences; Thierry Troosters, PhD, Study Chair — KU-Leuven, Faculty of Movement and Rehabilitation Sciences; Marc Decramer, PhD, Study Chair — University Hospital Leuven, Respiratory Division; Geert Verleden, PhD, Study Chair — University Hospital Leuven, Respiratory Division; Lieven Dupont, PhD, Study Chair — University Hospital Leuven, Respiratory Division
Locations (1):
- University Hospital Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Gutierrez-Arias R, Martinez-Zapata MJ, Gaete-Mahn MC, Osorio D, Bustos L, Melo Tanner J, Hidalgo R, Seron P. Exercise training for adult lung transplant recipients. Cochrane Database Syst Rev. 2021 Jul 20;7(7):CD012307. doi: 10.1002/14651858.CD012307.pub2. PMID 34282853